CLINICAL TRIAL: NCT06110221
Title: Oral Biofluid Levels of Activin-A and Interleukin-1 Beta Levels in Periodontal Health and Disease
Brief Title: Activin-A and Interleukin-1β Levels in Periodontitis
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Beral Afacan, Assoc. Prof., Aydin Adnan Menderes University
Other Study IDs: Activin-A
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Periodontitis; Gingivitis; Periodontal Health
MeSH Terms: conditions — Periodontitis; Gingivitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Periodontitis: This group consisted of patients with generalized stage III periodontitis, who had interproximal CAL≥5 mm and PD≥6 mm as well as radiographical bone loss extending to the mid-third of the root or beyond at 30% of the teeth or more. CAL was not caused by trauma-related gingival recession, dental caries extending into the cervical areas of the teeth, endodontic lesions draining through the marginal periodontium, and the distal bone loss in adjacent second molars due to extractions of third molars. They showed no more than four teeth loss due to periodontitis.
  Interventions: Other: Periodontal clinical measurements, GCF and saliva sampling
- Gingivitis: This group demonstrated no detectable interproximal CAL or radiographical bone loss. PD was ≤3 mm and BOP (%) was ≥30% in the entire mouth.
  Interventions: Other: Periodontal clinical measurements, GCF and saliva sampling
- Periodontal health: This healthy control group had an intact periodontium without detectable CAL and radiographical bone loss. PD was ≤3 mm and BOP (%) was <10% in the entire mouth.
  Interventions: Other: Periodontal clinical measurements, GCF and saliva sampling

INTERVENTIONS:
Other: Periodontal clinical measurements, GCF and saliva sampling — Clinical periodontal indices included probing depth (PD), clinical attachment loss (CAL), the dichotomous scoring of bleeding on probing (BOP +/-), gingival index (GI), and plaque index (PI). Clinical recordings were performed at six points (mesiobuccal, buccal, distobuccal, mesiopalatal, palatal, and distopalatal) of all teeth, except the 3rd molars.
  GCF and saliva samples were obtained 1 day following the clinical measurements. Unstimulated whole saliva was collected from all participants. GCF was sampled with paper strips from two deepest pockets in periodontitis group; the most inflamed sites with clinical signs of redness or edema in gingivitis group; and the sites without visible inflammation in periodontally healthy group. GCF and saliva samples were stored at -80 °C until further analysis.

SUMMARY:
Activin-A belongs to the transforming growth factor-beta superfamily and is a multifunctional cytokine that plays a role in inflammation, immune response, tissue repair and regeneration. Proinflammatory cytokine interleukin-1beta (IL-1β) can increase Activin-A expression in various cell types. This study aims to evaluate gingival crevicular fluid (GCF) and salivary Activin-A and IL-β levels in stage III periodontitis. Seventy-five systemically healthy and non-smoker volunteers consisting of 23 stage III periodontitis, 26 gingivitis and 26 periodontally healthy were enrolled. Full-mouth clinical periodontal indices were recorded, unstimulated whole saliva and GCF samples were obtained, Activin-A and IL-1β total amounts were determined by enzyme-linked immunosorbent assay. Statistical comparisons were performed using non-parametric tests.

DETAILED DESCRIPTION:
Participants were divided into three groups according to the diagnostic criteria proposed by the Classification of Periodontal and Peri-implant Diseases and Conditions; I. Periodontitis group (n=23), II. Gingivitis group (n=26) III. Periodontally healthy group (n=26)

Clinical periodontal indices included probing depth (PD), clinical attachment loss (CAL), the dichotomous scoring of bleeding on probing (BOP +/-), gingival index (GI), and plaque index (PI). Clinical recordings were performed at six points (mesiobuccal, buccal, distobuccal, mesiopalatal/mesiolingual, palatal/lingual, and distopalatal/distolingual) of all teeth, except the 3rd molars, by a single investigator using a conventional periodontal probe.

Interproximal radiographic bone loss on the digital panoramic radiographs were evaluated, as the ratio of the distance between the bone crest and the cemento-enamel junction to the length of the root.

GCF and unstimulated whole saliva samples were obtained 1 day following the clinical periodontal measurements. Immediately after saliva collection, GCF was collected from the buccal aspects of non-contiguous interproximal sites in two single-rooted teeth via steril paper strips. Fluid samples were obtained from two deepest pockets in periodontitis group and the most inflamed sites with clinical signs of redness or edema in gingivitis group. In the periodontally healthy groups, samples were taken from the sites without visible inflammation. All samples were stored at -80 °C until further analysis.

Measurement of Activin-A and IL-1β levels in GCF and saliva samples were performed by the commercially available enzyme-linked immunosorbent assay (ELISA) kits. While GCF cytokine levels were expressed as both total amounts at two samples per 30 s and concentrations, salivary cytokine levels were presented as concentrations.

A statistical software package was used for all data analyses. If the clinical and biochemical data did not present normal distribution as checked by Shapiro Wilk's normality test, the analyses were performed by using nonparametric methods. The Kruskal-Wallis test with Dunn-Bonferroni post hoc method was applied to compare the study groups regarding clinical indices and oral biofluid levels of Activin-A and IL-1β. The presence and degree of linear association of cytokine levels in GCF and saliva with clinical indices were analyzed by Spearman rank correlation coefficient. p<0.05 was considered as a threshold for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* the presence of no history of smoking (determined by self-reporting)
* at least 18 natural teeth excluding 3rd molars.

Exclusion Criteria:

* the presence of systemic conditions (diabetes mellitus, rheumatoid arthritis, cardiovascular system diseases, endocrine, immunologic, and mucocutaneous disorders) - use of antibiotics, antihypertensives immunosuppressive and anti-inflammatory drugs within the past 6 months and topical antiseptic solutions in the last 3 months
* having periodontal treatment in the previous year
* wearing removable partial dentures or orthodontic appliances
* restorative and endodontic therapy requirements
* pregnant or nursing women.

Ages: 27 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This prospective case-control study consecutively enrolled 75 individuals (39 females and 36 males and; aged 27 to 48 years; mean age, 37.30 ± 5.10 years) from the Department of Periodontology, School of Dentistry, Aydın Adnan Menderes University, Aydın, Turkey, in the period from March 2019 to January 2020.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
GCF Activin-A levels | 24 hours after clinical periodontal measurements
  total amount (ng)

CONTACTS AND LOCATIONS:
Overall Officials: Beral Afacan, Principal Investigator — Department of Periodontology, School of Dentistry, Aydın Adnan Menderes University
Locations (1):
- Aydın Adnan Menderes University, Aydin, Turkey (Türkiye)